CLINICAL TRIAL: NCT01899339
Title: Submassive Pulmonary Embolism Treatment With Ultrasound-Accelerated Thrombolysis
Brief Title: Long Term Effects of Treating Submassive Pulmonary Embolism With Ultra-sound Accelerated Thrombolysis
Acronym: SPEAR
Status: Completed | Type: Observational
Sponsor: Corewell Health West (Other)
Collaborators: EKOS Corporation (Industry)
Responsible Party: Principal Investigator, Michael F Knox, MD, Medical Doctor, Corewell Health West
Other Study IDs: 2013-069; Ekos (Other: spectrum health)
Record Dates: First submitted 2013-07-10; First posted 2013-07-15 (Estimated); Last update posted 2023-07-18 (Actual); Status verified 2023-07

CONDITIONS: Submassive Pulmonary Embolism
Keywords: submassive pulmonary embolism; Ultrasonic energy; Ekosonic Endovascular Device; RV:LV function after Pulmonary Embolism

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- pulmonary embolism: patients with submassive pulmonary embolism
  Interventions: Other: submassive PA treatment with Ekosonic endo device

INTERVENTIONS:
Other: submassive PA treatment with Ekosonic endo device — Ultra Sound energy along with tPA to treat submassive pulmonary embolism
  Other Names: Ekosonic Endovascular Device

SUMMARY:
Patients with Submassive Pulmonary Embolism treated with ultra-sound therapy will have an improved right ventricular function 72 hours post treatment.

ELIGIBILITY:
Inclusion Criteria:

* Patients with acute (< or = 14 days)symptomatic pulmonary embolism by CT Angiogram of the thorax with embolus involving at least one main or lower lobe pulmonary artery and RV:LV ratio > 0.9

Exclusion Criteria:

* age > 80
* Recent thrombolytic therapy (with in 4 days)
* Active bleeding or know bleeding diathesis
* Known coagulopathy (including treatment with vitamin K antagonists) INR > 3 and/or PTT > 50
* Thrombocytopenia (PLT cound < 100,000)
* History of any intracranial or intraspinal surgery, trauma or bleed
* Intracranial neoplasms, AVM, or aneurysm
* Recent (< 1 month) GI bleed
* Recent (< 3 months) internal eye surgery or hemorrhagic retinopathy
* Recent (< 7 days) major surgery, trauma, or obstetrical delivery
* Renal insufficiency with eGFR < 45 ml/min
* Known allergy, hypersensitivity, or thrombocytopenia from heparin or tPA
* Hemodynamic instability defined as need for cardiopulmonay resuscitation, Systolic BP > 90 mm Hg for > 15 min or need for pressor agents to maintain BP > 90.
* Severe Hypertension (sustained systolic > 180 mm Hg or diastolic > 90 mm Hg.
* Pregnant patients
* known right to left shunt
* Large (>10 mm)intracardiac thrombus
* Use of thrombolytics or glycoprotein IIb/IIIa antangonists within 3 days of inclusion.
* Life expectancy < 30 days

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All patient presenting to the Emergency Department with submassive pulmonary hypertension over the age of 18.
Sampling Method: Probability Sample
Enrollment: 25 (Actual)
Dates: Start 2013-05; Primary Completion 2019-02 (Actual); Study Completion 2019-02 (Actual)

PRIMARY OUTCOMES:
Change in Right Ventricular:Left Ventricular ratio | baseline to 72 hours post
  Treatment will show improved Right Ventricular:Left Ventricular ratio at 72 hours post.

SECONDARY OUTCOMES:
recurrent pulmonary embolism | 30 days post procedure
  Will assess whether a recurrent Pulmonary Embolism has happened at 30 day post procedure or earlier

CONTACTS AND LOCATIONS:
Overall Officials: Michael Knox, MD, Principal Investigator — Spectrum Health Hosptials and ARS
Locations (1):
- Spectrum Health Hospitals, Grand Rapids, Michigan, United States